CLINICAL TRIAL: NCT06437730
Title: Comparison of Integrated Neuromuscular Inhibition Technique and Dry Needling on Trigger Points in Patient With Knee Osteoarthritis
Brief Title: Comparison of INIT and Dry Needling on Trigger Points in Knee OA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Iqra Iftikhar
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
Keywords: Trigger Points,; Knee Osteoarthritis,; Dry Needling,; Integrated Neuromuscular Inhibition Technique,
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group: 1 (Experimental): MTrPs points will be released with ischemic compression, position of ease will be acquired, and in the last METs will be performed. Ischemic compression applied through thumb on trigger point present in any muscle around the knee joint.
  Interventions: Other: Integrated Neuromuscular Inhibition Technique:
- Group: 2 (Experimental): Dry needle will be targeting trigger points (TrPs) using in-and-out techniques such as 'pistoning' or 'sparrow pecking'. 0.25x25mm needle is inserted.
  Interventions: Other: Dry needling:

INTERVENTIONS:
Other: Integrated Neuromuscular Inhibition Technique: — MTrPs points will be released with ischemic compression, position of ease will be acquired, and in the last METs will be performed. Ischemic compression applied through thumb on trigger point present in any muscle around the knee joint. Compression will be increased gradually until first resistance will feel and maintained until it resolves, further increases then until no tissue resistance will be felt under thumb. This process is maintained for 30sec and repeated 3-5 times per session. Positional release technique: after applying pressure on trigger point, patient will acquire position of ease that is maintained for 20 sec whether its extension or flexion of knee. This process is repeated 3-5 times per session. Muscle Energy Technique will be applied on the muscle in which isometric contraction is maintained for 7-10sec against 20-25% strength. After completion of muscular contraction, the limb is moved away for muscular stretch and then position is maintained for 30 seconds
  Arms: Group: 1
Other: Dry needling: — Dry needle will be targeting trigger points (TrPs) using in-and-out techniques such as 'pistoning' or 'sparrow pecking'. 0.25x25mm needle is inserted.
  For vastus laterals patient is supine line with knee extended performing an isometric quadriceps contraction, maintaining a clean technique by using gloves and performing an alcohol wipe down bracket the tissue to be treated and inserting needle with direct approach towards the femur, performing pistoning. For vastus medialis patient is supine line with 30 degrees of knee flexion. A headless 0.25x25mm needle fixed between the fingers of non-dominant hand and inserted perpendicularly to the MTrPs with metacarpophalangeal flexion extension of 1st and 2nd fingers of dominant hand. For Gastrocnemius patient is prone lying and bolstered supported slight knee bend, for the upper part anterior medial approach is used and center of muscle belly slight medial anterior approach is used.
  Arms: Group: 2

SUMMARY:
The purpose of the study is to compare the effects of Integrated Neuromuscular Inhibition Technique and Dry Needling on Functional Disability, Pain and Range of Motion. A randomized control trial will be conducted at Wah General Hospital Taxila. The sample size is 36 calculated through G-Power but I recruited 50. The participants were divided into two interventional groups each having 18 participants. Tools used in this study are Goniometer, NPRS, WOMAC, and Self structured Questionnaire. Data will be collected before and immediately after the application of interventions. Data will be analyzed through SPSS.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is also known as degenerative joint disease, in which there is progressive loss of articular cartilage due to wear and tear. Knee osteoarthritis can be classified into two types, primary and secondary. Primary osteoarthritis is defined as degeneration of articular cartilage without any underlying cause. Secondary osteoarthritis can be caused due to either an abnormal amount of forces placed across the joint in a result of post-traumatic cause or due to abnormal articular cartilage, for example Rheumatoid arthritis. The prevalence of knee OA is higher as compared to other types of OA. As with increasing age and longer lifetime and higher average weight of population the incidence of knee OA increases, particularly in obese women. Women have a greater prevalence (42.1%) than do men (31.2%). There are different grades of knee OA. In Grade 1 There is a swelling of articular cartilage along with mild fibrillation in superficial zone. In Grade 2 Small portion of cartilage is lost and fibrillation occurs in deeper zone and clusters of chondrocytes begun to form. In Grade 3 formation of chondrons occurs and vertical fissures have advanced into middle zone. Early OA changes affects the superficial and middle zone of cartilage. There are different risk factors for developing Knee OA that includes age, Female Gender, Menopause, heredity, repetitive micro and macro trauma, alcohol and tobacco use and joint surgery. Some risk factors are modifiable and some are non-modifiable. Modifiable factors include: any trauma, occupation, weight, muscle weakness or imbalance, Prolonged standing and repetitive knee bending. Non-modifiable risk factors include Gender - females, Age, Genetics and Race. There can be different causes of knee OA including family history, obesity, age, diabetes, systemic inflammatory mediators, lower limb alignment, trauma and inflammation by metabolic syndrome. Diagnosis of Knee OA is mainly based on symptoms and X-rays according to Kellgren and Lawrence system for classification of Osteoarthritis. The Knee OA most common symptom is pain around knee joint, Pain can be of different nature such as dull, intermittent or sharp. Pain intensity can also vary from mild to moderate to severe. The Range of motion can also be decreased in knee OA. Other symptoms include grinding and popping sounds. Swelling, locking and giving way of the knee can also be seen in later stages. Inconsistencies are observed, in which they explain presence of Myofascial trigger points in surrounding muscles around knee. Studies showed treatment of trigger points will cause reduction in pain and improvement in functional capacity in Knee OA patients. There are different techniques to treat trigger points e.g. Dry needling and Integrated neuromuscular inhibition technique.

Study reported that there's significant reduction in pain and disability along with improved ROM in Knee Osteoarthritis patients who received Integrated Neuromuscular Inhibition Technique combined with Conventional treatment.

Another study conducted on Effect of Integrated Neuromuscular Inhibition Technique on Iliotibial Band Tightness in Osteoarthritis of Knee and their study concluded that there is a significant effect of Integrated Neuromuscular Inhibition Technique on iliotibial band tightness in osteoarthritis of knee.

Study was done to check effect of Dry needling in an exercise program for older adults with knee OA, The study concluded Despite the pain intensity and disability clinically relevant improvement for both DN and Sham-DN combined with exercise, 6 sessions of DN added to a therapeutic exercise program for older adults with KO did not seem to improve pain intensity and functionality.

Study conducted on Dry needling versus INIT on upper trapezius myofascial trigger points. According to study findings DN was more effective than INIT on management of upper trapezius active myofascial trigger points.

Proper evidence behind comparative effect of INIT and DN on trigger points in knee OA patient is sparse and there are less number of studies with limited methodological design on these techniques. This study will contribute to compare the ef-fects of INIT and Dry Needling on Functional Disability, Pain and ROM in patients with knee OA, and to check whether which technique is more effective in treating trigger points in Knee Osteoarthritis patients

ELIGIBILITY:
Inclusion Criteria:

Osteoarthritis Grade-1 to 2 Positive jump sign Vastus medialis(75.43%), Vastus laterals(65.78%), Gastrocnemius

Exclusion Criteria:

* Patient with history of RA or any autoimmune disorder Any systematic Illness Patient with Varicose vein Post traumatic, Post-Surgical and Post fractured

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index | 6th day
  The WOMAC pain score is a numerical score that measures pain, stiffness, and functional limitations. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for pain, 0-8 for stiffness, and 0-68 for physical function.
Numeric Pain Rating Scale | 6th day
  The numeric pain rating scale is a scale for self-report of pain intensity. It is an 11-point scale, where 0 means no pain and 10 means the worst possible pain.
Goniometer: | 6th day
  A goniometer is a device used in physical therapy to measure a joint's range of motion. It is essentially a protractor with two arms extending from it, used to measure a joint's range of motion.. There are two "arms" one that is stationary and one that is movable-that are hinged together. Each is positioned at specific points on the body with the center of the goniometer aligned at the joint of interest. The goniometer can be used to measure many joints such as the knee, hip, shoulder, or wrist.
Kellgren and Lawrence system for classification of Osteoarthritis: | 6th day
  It is a common method of classifying the severity of Osteoarthritis using five grades
  The grades are as follows:
  Grade 0 (none): definite absence of x-ray changes of osteoarthritis Grade 1 (doubtful): doubtful joint space narrowing and possible osteophytic lipping Grade 2 (minimal): definite osteophytes and possible joint space narrowing Grade 3 (moderate): moderate multiple osteophytes, definite narrowing of joint space and some sclerosis and possible deformity of bone ends Grade 4 (severe): large osteophytes, marked narrowing of joint space, severe sclerosis and definite deformity of bone ends.

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScPT, Principal Investigator — Riphah International University
Locations (1):
- Wah General Hospital,, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsu H, Siwiec RM. Knee Osteoarthritis. 2023 Jun 26. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507884/ PMID 29939661
- [Background] Lespasio MJ, Piuzzi NS, Husni ME, Muschler GF, Guarino A, Mont MA. Knee Osteoarthritis: A Primer. Perm J. 2017;21:16-183. doi: 10.7812/TPP/16-183. PMID 29035179
- [Background] Heidari B. Knee osteoarthritis diagnosis, treatment and associated factors of progression: part II. Caspian J Intern Med. 2011 Summer;2(3):249-55. PMID 24049581
- [Background] Favero M, Ramonda R, Goldring MB, Goldring SR, Punzi L. Early knee osteoarthritis. RMD Open. 2015 Aug 15;1(Suppl 1):e000062. doi: 10.1136/rmdopen-2015-000062. eCollection 2015. PMID 26557380
- [Background] Ejaz F, Safdar M, Ejaz H. Comparative Effectiveness of Integrated Neuromuscular Inhibition Technique Along with Conventional Treatment Vs Conventional Treatment Alone in Patients of Knee Osteoarthritis. Pakistan Journal of Medical & Health Sciences. 2023;17(01):859-.
- [Background] Albin SR, Koppenhaver SL, MacDonald CW, Capoccia S, Ngo D, Phippen S, Pineda R, Wendlandt A, Hoffman LR. The effect of dry needling on gastrocnemius muscle stiffness and strength in participants with latent trigger points. J Electromyogr Kinesiol. 2020 Dec;55:102479. doi: 10.1016/j.jelekin.2020.102479. Epub 2020 Oct 9. PMID 33075711
- [Background] Muraja S, Markulinčić B. FRI0597-HPR The effect of physical therapy on functional status and synovial perfusion in patients with knee osteoarthritis. Annals of the Rheumatic Diseases. 2013;72(Suppl 3):A578-A.
- [Background] Mayoral O, Salvat I, Martin MT, Martin S, Santiago J, Cotarelo J, Rodriguez C. Efficacy of myofascial trigger point dry needling in the prevention of pain after total knee arthroplasty: a randomized, double-blinded, placebo-controlled trial. Evid Based Complement Alternat Med. 2013;2013:694941. doi: 10.1155/2013/694941. Epub 2013 Mar 27. PMID 23606888
- [Background] Chavan SE, Shinde S. Effect of Integrated Neuromuscular Inhibition Technique on Iliotibial Band Tightness in Osteoarthritis of Knee
- [Background] Sanchez-Romero EA, Pecos-Martin D, Calvo-Lobo C, Ochoa-Saez V, Burgos-Caballero V, Fernandez-Carnero J. Effects of dry needling in an exercise program for older adults with knee osteoarthritis: A pilot clinical trial. Medicine (Baltimore). 2018 Jun;97(26):e11255. doi: 10.1097/MD.0000000000011255. PMID 29952993
- [Background] Abdelaziz YM, Abulkasem ST, Yamny AA. Dry Needling Versus Integrated Neuromuscular Inhibition Technique on Upper Trapezius Myofascial Trigger Points. Egypt J Appl Sci. 2020;35:45-56.